CLINICAL TRIAL: NCT04752657
Title: eFramingham Heart Study Randomized Controlled Trial #2
Brief Title: Second eFramngham Heart Study
Acronym: eFHS-2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: H-40737; 5R01HL141434-03 (NIH)
Record Dates: First submitted 2021-02-09; First posted 2021-02-12 (Actual); Results first posted 2025-03-19 (Actual); Last update posted 2025-03-19 (Actual); Status verified 2025-02

CONDITIONS: Cardiovascular Diseases
Keywords: Framingham Heart Sudy; eFHS; mhealth; patient provider communication; user engagement
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Intervention Model Description: Each participant will be randomized to one of the 2 groups. A statistician will generate randomization lists with the use of randomly permuted blocks of varying sizes, with stratification according to participant's age (≤75 years vs. >75 years) and type of phone (android vs. iphone). Randomization will be implemented centrally through the app.
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): The experimental group will receive the physical function survey at weeks 2, 10, 18, and 26; the physical activity survey at weeks 2, 14, and 26; the events survey at weeks 2, 6, 10, 14, 18, 22, and 26. The administration of the cognition, pain, mood, and psychosocial surveys follow the same pattern for both groups.
  Interventions: Other: Delayed administration of survey modules
- Control Group (Active Comparator): The control group will receive the physical function survey at weeks 0, 8, 16, and 24; the physical activity survey at weeks 0, 12, and 24; the events survey at weeks 0, 4, 8, 12, 16, 20, and 24. The administration of the cognition, pain, mood, and psychosocial surveys follow the same pattern for both groups.
  Interventions: Other: Regular administration of survey modules

INTERVENTIONS:
Other: Delayed administration of survey modules — The intervention consists in delaying the administration of the physical function, physical activity, and events survey modules by 2 weeks
  Arms: Experimental Group
Other: Regular administration of survey modules — The physical function, physical activity, and events survey modules are administered according to the regular pattern
  Arms: Control Group

SUMMARY:
In the electronic Framingham Heart Study (eFHS), the investigators developed and deployed a mobile app to collect cardiovascular risk factors and event data and test them against cardiovascular data collected in the Framingham research clinic for the FHS.

Participants enrolled in eFHS receive a series of digital surveys modules to complete on a regularly occurring schedule. The objective of the planned randomized trial is to test the effect of administering half of survey modules every 2 weeks versus all survey modules every 4 weeks on improving participants' response rates.

There will be 4 survey periods. Period 1 encompasses all survey modules administered from baseline up to week 8 (19 surveys/tasks per participant); period 2 from week 8 up to week 16 (18 surveys/tasks per participant); period 3 from week 16 up to week 24; period 4 from week 24 (16 surveys/tasks per participant).

DETAILED DESCRIPTION:
Participants in eFHS are invited to enroll from the FHS Offspring and Omni Group 1 Cohorts during the in-person examination 10/5 at the FHS Research Center in Framingham, Massachusetts (MA), USA or remotely from home after the in-person examination. All eFHS participants have the eFHS myDataHelps mobile app (developed by FHS investigators with CareEvolution our industry partner) installed on their smartphone. The eFHS app allows communication with participants through notifications and data collection. Participants are asked to answer health surveys administered through the app.

Survey assessments will include 6 modules: cognition, pain, mood, physical function and performance, physical activity, and events. The interventions are defined by the patterns of administration of survey modules to the experimental and control groups. The administration of the cognition, pain, mood, and psychosocial modules follow the same pattern for both groups. However, the administration of the physical function, physical activity, and events modules is delayed by 2 weeks in the experimental group as compared to the control group.

ELIGIBILITY:
Inclusion Criteria:

* Invited to enroll from the FHS Offspring and Omni Group 1 Cohorts during the in-person examination 10/5 at the FHS Research Center
* English speaking
* English language reading proficiency
* Owns an iPhone with compatible iOS (version 10.0 or higher) or Android (version 5.0 or higher)
* Residence in the United States
* Provision of permissions for notifications and data sharing with the Research Center
* Provision of signed and dated informed consent (within the eFHS mobile app)

Exclusion Criteria:

* Limited and non-readers

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 492 (Actual)
Dates: Start 2021-06-21 (Actual); Primary Completion 2023-12-28 (Actual); Study Completion 2023-12-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joanne Murabito, Principal Investigator — Framingham Heart Study
Locations (1):
- Framingham Heart Study, Framingham, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
The datasets generated and analyzed during this study are available from the research team upon reasonable request.
Supporting Information: Study Protocol, SAP
Time Frame: Investigators can research out to the research team from time of publication.
Access Criteria: The data will be accessible from the research team via FHS guidelines at https://www.framinghamheartstudy.org/fhs-for-researchers/data-available-overview/

REFERENCES:
- [Derived] Zhang Y, Rong J, Wang X, Schramm E, Pathiravasan CH, Borrelli B, Faro JM, Benjamin EJ, Trinquart L, Liu C, Murabito JM. Smartphone App-Based Survey Deployment Patterns and Longitudinal Response Rate: Randomized Controlled Trial. J Med Internet Res. 2025 Oct 10;27:e73972. doi: 10.2196/73972. PMID 41071587

RESULTS

PARTICIPANT FLOW:
Groups:
- Experimental- Two-week Group: Delayed administration of the physical function, physical activity, and events survey modules by 2 weeks.
- Control- Four-week Group: The physical function, physical activity, and events survey modules are administered according to the regular 4-week pattern.
Period: Period 1- Baseline up to Week 8
Arm/Group | Experimental- Two-week Group | Control- Four-week Group
Started | 248 | 244
Completed | 248 | 244
Not Completed | 0 | 0
Period: Period 2- Week 8 up to Week 16
Arm/Group | Experimental- Two-week Group | Control- Four-week Group
Started | 248 | 244
Completed | 248 | 244
Not Completed | 0 | 0
Period: Period 3- Week 16 up to Week 24
Arm/Group | Experimental- Two-week Group | Control- Four-week Group
Started | 248 | 244
Completed | 248 | 244
Not Completed | 0 | 0
Period: Period 4- Week 24 to Study Completion
Arm/Group | Experimental- Two-week Group | Control- Four-week Group
Started | 248 | 244
Completed | 248 | 244
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Experimental- Two-week Group | Control- Four-week Group | Total
Number analyzed (Participants) | 248 | 244 | 492
Age, Continuous [Mean (Standard Deviation); unit: years] | 74.0 (6.2) | 73.9 (6.3) | 73.9 (6.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 148 | 136 | 284
  Male | 100 | 108 | 208
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 209 | 205 | 414
  Other | 39 | 39 | 78
Region of Enrollment [Number; unit: participants]
  United States | 248 | 244 | 492

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Surveys/Tasks Returned in Period 1
Description: Proportion of surveys/task returned per participant (partially or fully completed) from baseline, up to week 8, will be documented on the eFHS app.
Time Frame: baseline, up to week 8
Measure: Mean (Standard Deviation); unit: proportion of surveys returned
Arm/Group | Experimental- Two-week Group | Control- Four-week Group
Number analyzed (Participants) | 248 | 244
proportion of surveys returned | 0.85 (0.28) | 0.85 (0.29)

2. Primary Outcome: Proportion of Surveys/Tasks Returned in Period 2
Description: Proportion of surveys/task returned per participant (partially or fully completed) from week 8, up to week 16, will be documented on the eFHS app.
Time Frame: week 8, up to week 16
Measure: Mean (Standard Deviation); unit: proportion of surveys returned
Arm/Group | Experimental- Two-week Group | Control- Four-week Group
Number analyzed (Participants) | 248 | 244
proportion of surveys returned | 0.75 (0.40) | 0.72 (0.42)

3. Primary Outcome: Proportion of Surveys/Tasks Returned in Period 3
Description: Proportion of surveys/task returned per participant (partially or fully completed) week 16, up to week 24, will be documented on the eFHS app.
Time Frame: week 16, up to week 24
Measure: Mean (Standard Deviation); unit: proportion of surveys returned
Arm/Group | Experimental- Two-week Group | Control- Four-week Group
Number analyzed (Participants) | 248 | 244
proportion of surveys returned | 0.71 (0.43) | 0.67 (0.45)

4. Primary Outcome: Proportion of Surveys/Tasks Returned in Period 4
Description: Proportion of surveys/task returned per participant (partially or fully completed) week 24, to completion of study usually 26 weeks, will be documented on the eFHS app.
Time Frame: week 24, to completion of study usually 26 weeks
Measure: Mean (Standard Deviation); unit: proportion of surveys returned
Arm/Group | Experimental- Two-week Group | Control- Four-week Group
Number analyzed (Participants) | 248 | 244
proportion of surveys returned | 0.66 (0.44) | 0.59 (0.47)

5. Secondary Outcome: Proportion of Questions/Task Completed Per Participant in Period 1
Description: Proportion of questions/task completed per participant from all survey modules administered from baseline to week 8, will be documented on the eFHS app.
Time Frame: baseline, up to week 8
Measure: Mean (Standard Deviation); unit: proportion of questions completed
Arm/Group | Experimental- Two-week Group | Control- Four-week Group
Number analyzed (Participants) | 248 | 244
proportion of questions completed | 0.86 (0.28) | 0.88 (0.29)

6. Secondary Outcome: Proportion of Questions/Task Completed Per Participant in Period 2
Description: Proportion of questions/task completed per participant from week 8 to week 16, will be documented on the eFHS app.
Time Frame: week 8, up to week 16
Measure: Mean (Standard Deviation); unit: proportion of questions completed
Arm/Group | Experimental- Two-week Group | Control- Four-week Group
Number analyzed (Participants) | 248 | 244
proportion of questions completed | 0.77 (0.40) | 0.74 (0.42)

7. Secondary Outcome: Proportion of Questions/Task Completed Per Participant in Period 3
Description: Proportion of questions/task completed per participant from week 16 to week 24, will be documented on the eFHS app.
Time Frame: week 16, up to week 24
Measure: Mean (Standard Deviation); unit: proportion of questions completed
Arm/Group | Experimental- Two-week Group | Control- Four-week Group
Number analyzed (Participants) | 248 | 244
proportion of questions completed | 0.73 (0.43) | 0.70 (0.45)

8. Secondary Outcome: Proportion of Questions/Task Completed Per Participant in Period 4
Description: Proportion of questions/task completed per participant from week 24 to study completion, will be documented on the eFHS app.
Time Frame: week 24, to completion of study usually 26 weeks
Measure: Mean (Standard Deviation); unit: proportion of questions completed
Arm/Group | Experimental- Two-week Group | Control- Four-week Group
Number analyzed (Participants) | 248 | 244
proportion of questions completed | 0.68 (0.44) | 0.61 (0.47)

ADVERSE EVENTS:
Time Frame: 26 weeks
Arm/Group | Experimental- Two-week Group | Control- Four-week Group
All-Cause Mortality (participants affected / at risk) | 0/248 | 0/244
Serious Adverse Events (participants affected / at risk) | 0/248 | 0/244
Other Adverse Events (participants affected / at risk) | 0/248 | 0/244

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-10-01): https://cdn.clinicaltrials.gov/large-docs/57/NCT04752657/Prot_SAP_000.pdf
  • Informed Consent Form (2021-05-28): https://cdn.clinicaltrials.gov/large-docs/57/NCT04752657/ICF_001.pdf